CLINICAL TRIAL: NCT05775978
Title: Testing the Effects of Two Psycho-educational Programs on Well Being and Academic Performance of Undergraduate Students at the University of Granada (Spain): An Interventional Study
Brief Title: Psycho-educational Training in Undergraduate Students at the University of Granada (Spain). Second Edition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercedes García de Quesada (Other)
Collaborators: Cívitas-UGR Chair: Sustainability, Innovation and Development, Granada, Spain (Unknown)
Responsible Party: Sponsor-Investigator, Mercedes García de Quesada, Principal Investigator, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Cívitas-UGR 2023
Record Dates: First submitted 2023-02-25; First posted 2023-03-20 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Empathy; Compassion; Attention; Psychological Distress; Life Stress; Anxiety; Creativity; Emotional Intelligence
Keywords: Sustainable Development; Mindfulness; Curriculum Design; Cognitive Behavioral Training; Learning in Higher Education; Employability
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Students are randomly assigned to three groups: the MBSR group that receives an adapted version of the MBSR program, the Más Presente group that receives training on transversal competences following the EU framework, LifeComp, and a third group that receives a neuro-muscular stimulation-based program. All participants are asked to fill in an informed consent and a demographic questionnaire to determine eligibility. Eligible participants are randomly assigned to either group. The three programs are given simultaneously.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator: researchers have no information on participants' allocation in the groups; a research assistant from the Cognitive Neuroscience Group of the CIMCYC is designated for this purpose. None of the participants are students of any of the researchers. For the purpose of communicating with the participants over group allocation, another lecturer from the UGR is appointed. Outcome Assessors: all measures are collected online via the UGR LimeSurvey platform and no recording of group assignment is introduced in the system. Care providers: they are not informed about the outcome measures or specific research hypothesis regarding expected effects for each program. Participants: although it is not possible to blind their assignment to the groups in this type of study, they are not informed about the specific hypothesis regarding the expected outcomes of the programs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UGRComp group (Experimental): This arm will instruct the students on the Más Presente program. This is a socio-emotional competence-based program which has been designed following the European LifeComp framework. This program is a combination of theory and practice aimed at developing the core elements of personal, social and learning to learn key competences for lifelong learning.
  Interventions: Behavioral: Más Presente, the UGRComp program
- MBSR group (Experimental): This arm will instruct the students on the Mindfulness-Based Stress Reduction (MBSR) program. The MBSR is a secular, evidence-based practice originally developed for chronic pain, but which has reported positive results among an array of clinical and nonclinical populations. This program aims to cultivate non-judgmental attention to and awareness of present moment experience while promoting stress reduction.
  Interventions: Behavioral: The MBSR program
- Neuro-muscular stimulation group (Active Comparator): The students in this arm will receive training on physical wellbeing and neuro-muscular stimulation.
  Non-specific factors such as number and duration of sessions, or instructor training and qualifications will match the other 2 experimental groups. Active ingredients such as mindfulness or socio-emotional training are not contained in the program.
  Interventions: Behavioral: Neuro-muscular stimulation

INTERVENTIONS:
Behavioral: Más Presente, the UGRComp program — Más Presente, the UGRComp program is based upon the European LifeComp framework (Sala, Punie, Garkov and Cabrera Giraldez 2020) and covers intra and interpersonal, emotional, cognitive and metacognitive aspects. Created at the University of Granada by an interdisciplinary group of experts, it focuses on three core elements (self-regulation, empathy and growth mindset) as they are the pre-requisites for developing all other elements across framework areas. It consists of 8 weekly classes, 2 hours each, together with a day of intensive practice. The program is structured along the following topics: The Underpinnings of Más Presente; Awareness and Concentration: our Body; Managing our Emotional Laberynth; Walking with Directionality, Sense and Conscience; Empathy, Presence and Connection; Empathic Listening and Honest Expression: Non-violent communication; Growth Mindset, Creativity and Divergent Thinking; And Now what? The First Day of the Rest of My Life.
  Other Names: The EU socio-emotional based program adapted to the UGR context
  Arms: UGRComp group
Behavioral: The MBSR program — The MBSR program is a group-based therapy which teaches mindfulness skills through a range of formal and informal mindfulness practices. Created by Kabat-Zinn (1982), in the current study it is taught by an officially accredited instructor and is compliant with the guidelines established by Brown University and the University of Massachusetts, USA. It originally consists of 8 weekly classes, 2 hours each (18 hours direct instruction), together with a day of intensive practice. The program is structured along the following topics: The Underpinnings of MBSR; The Perception of Reality; Power in Being Present; Understanding Stress: The Mind-Body Relation; Responding to Stress; Communication and Personal Relations; Daily Life Management; My Personal Plan: "What lies ahead".
  Other Names: Mindfulness-Based Stress Reduction program
  Arms: MBSR group
Behavioral: Neuro-muscular stimulation — Subjects will receive weekly sessions with a combination of educational sessions and specific physical exercises to enhance physical wellbeing and prevent neuro-degeneration . After spotting the therapeutic targets for each subject, a 4-phase program will be designed for each subject aimed at improving lifestyle habits and general wellbeing.
  Arms: Neuro-muscular stimulation group

SUMMARY:
The new professional profiles highlight the need to incorporate competences such as self-regulation, communication or growth mindset in the academia. Not only is this important for employability; a step further is needed. It's necessary to equip learners with knowledge, skills and attitudes that help them become agents of change and shape sustainable futures in our current complex society.

Within the framework of an agreement signed between the University of Granada (UGR), Spain, and, one of the leading real state firms in Spain, Cívitas, a course and a parallel study have been launched that will provide research and training in these competences at a degree level. It is part of the Sustainable Human Development Training Pathway of the Vice-Rectorate for Equality, Inclusion and Sustainability.

The main objective of the study is to test whether participating in a competence-based course can improve students' cognitive, emotional and personal traits as well as academic performance. Together with this main purpose, the present study also aims to compare the effects of two competence-based programs on the students' ability to improve specific aspects of cognition, emotional intelligence, creativity or academic performance among others. Both programs involve training sustained attention and an accepting and open attitude though they differ in several aspects of their methods, intention and aims.

Drawing conclusions from the research and outcomes, pedagogies which are best suited to develop theses competences at the Higher Education level will be suggested. Assessment and certification of this kind of competences will also be proposed.

DETAILED DESCRIPTION:
The content of the UGRComp program (Más Presente, Arm 1) was designed in 2021 using the European LifeComp framework, the content of the Mindfulness-Based Stress Reduction program (MBSR, Arm 2) follows the University of Massachusetts and Brown University specifications, and the content of the neuro-muscular stimulation program has been designed for the purpose of this study and is a combination of educational sessions and specific physical exercises to enhance physical wellbeing and prevent neuro-degeneration (Arm 3). Arms 1 and 2 will attend classes at the University of Granada premises. Arm 3 will receive training in neuro-muscular stimulation.

Instructors of the three arms are fully certified and have more than 10 years of professional experience in the field. All UGR undergraduate students are informed and invited to participate both in the course and in the study. They can choose to participate either in the study alone, in the course alone or in both. However, they are advised that, in the event that there are more applications than places, priority will be given to those who have registered earlier and those who choose to do the study.

So that the 3 ECTS credits of the course can be validated, the petition was inserted in a broader proposal by the Vice-Rectorate for Equality, Inclusion and Sustainability as part of the Sustainable Human Development Training Pathway. In this petition, the content of the course, design and aim of the study, potential participants, duration and other issues related with the project were included and explained.

The UGR grants some facilities (lecture rooms and Administrative and Support Staff's help). Vice-Rectorate for Equality, Inclusion and Sustainability will be responsible of the accreditation and certification processes. The Civitas-UGR Chair is responsible of co-funding and the study members from the Mind, Brain and Behaviour Research Center (CIMCYC) of the University of Granada (Spain) are responsible of study design, LimeSurvey management, randomization and data analysis.

All participants are asked to fill in an informed consent, a demographic questionnaire to determine eligibility and a battery of tests. Eligible participants are randomly assigned to either group.

All questionnaires are uploaded to the UGR LimeSuvey platform, an open source online survey tool specially designed to develop, publish and collect survey responses. This software is the one recommended by the University of Granada to present and collect online data for research purposes as it complies with all current legislation and ensures that all protection data requirements are being effectively met.

For specific security guarantees, an institutional email account is used through which all communication related to the project is carried out. In the same line, all the documentation generated within the project is uploaded and shared on a virtual cloud owned by the UGR (www.ugrdrive.ugr.es). It is expected to find improvements in all measures (psychological and academic) in the two experimental groups (students in Arms 1 and 2) after completing the course compared to pre-training and compared to an active control group (students in Arm 3). In order to measure potential specific effects of each mindfulness program, pre-training to post-training psychological measures will be compared once completed the program. Altogether, this applied study might help to elucidate whether these important transversal competences and soft skills can improve with mindfulness-based techniques and ultimately could be recommended as part of the official curricula of degree in Higher Education.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled at the University of Granada, Spain. Bachelor's Degree level

Exclusion Criteria:

* Current psychotherapy or history of psychotic disorder or neurological condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Change on the Spanish Short Self-Regulation Questionnaire (SSSRQ) | Baseline, 4 months
  17 items self-report scale, translated and validated into Spanish, that measures cognitive and behavioural aspects of self-regulation (Garzón et al. 2017). Respondents rate a series of statements on a 5-point Likert scale, with 1 being "strongly disagree" and 5 being "strongly agree"
Change on Guilford's Alternative Uses Test (GAU) | Baseline, 4 months
  Scoring in terms of originality, fluency, elaboration and flexibility. The higher the score the better the creativity and divergent thinking.
Change on the Five Facets Mindfulness Questionnaire (FFMQ) | Baseline, 4 months
  A 39-item self-report scale, translated and validated into Spanish, that measures mindfulness traits (Baer et al 2006, 2010; Cebolla et al 2012). Respondents rate a series of statements on a 5-point Likert scale, with 1 being "never" and 5 being "very often".
Change on the Depression Anxiety Stress Scale (DASS) | Baseline, 4 months
  A 21-item self-report scale, translated and validated into Spanish, that measures depression, anxiety and stress levels (Henry and Crawford 2005, Bados et al. 2005). Respondents rate a series of statements on a 4-point Likert scale, with 0 being "not at all true of me" and 3 being "very true of me".
Change on the Mind Wandering questionnaire (MW) | Baseline, 4 months
  An 8-item self-report scale, translated and validated into Spanish, that measures the levels of the mind wandering trait (Carriere et al. 2013). Respondents rate a series of statements on a 7-point Likert scale, with 1 being "almost never" and 7 being "almost always".
Change on the Basic Empathy Scale (BES) | Baseline, 4 months
  A 20-item self-report scale, translated and validated into Spanish, that measures affective and cognitive empathy (Villadangos et al. 2016). Respondents rate a series of statements on a 5-point Likert scale, with 1 being "strongly disagree" and 5 being "strongly agree".

SECONDARY OUTCOMES:
Academic qualifications extracted from the subjects' undergraduate transcript | Up to 4 years
  Results from primary outcome are associated with academic performance of students' core subjects.
Qualitative questionnaire on students' experience | 4 months
  This qualitative questionnaire with open ended questions builds directly on the results from the quantitative phase. The quantitative results are interpreted in more detail through the qualitative data.
Concentration of participants | Baseline, 4 months
  Every two questionnaires a control question will be inserted in order to test internal validity.
Eysenck Personality Inventory (EPI) | Baseline, 4 months
  A 24-item self-report scale to assess neuroticism and social conformity and desirability. Respondents rate a series of statements on a yes/no scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes T. García de Quesada, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Spain

REFERENCES:
- [Background] Sala A, Punie Y, Garkov V, Cabrera Giraldez M. LifeComp: The European framework for personal, social, and learning to learn key competence. Publications Office of the European Union. 2020.
- [Background] Baer RA, Samuel DB, Lykins EL. Differential item functioning on the Five Facet Mindfulness Questionnaire is minimal in demographically matched meditators and nonmeditators. Assessment. 2011 Mar;18(1):3-10. doi: 10.1177/1073191110392498. Epub 2010 Dec 30. PMID 21193491
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Cabello R, Salguero JM, Fernández-Berrocal P, Gross JJ. A Spanish adaptation of the emotion regulation questionnaire. Eur J Psychol Assess [Internet]. 2013; 29(4): 234-40. Available from: www.scopus.com
- [Background] Cebolla A, García-Palacios A, Soler J, Guillen V, Baños R, Botella C. Psychometric properties of the Spanish validation of the Five Facets of Mindfulness Questionnaire (FFMQ). The European Journal of Psychiatry. 2012; 26(2): 118-126.
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Bados A, Solanas A. Andrés R. Psychometric properties of the Spanish version of Depression, Anxiety and Stress Scales (DASS). Psicothema. 2005; 17(4): 679-683.
- [Background] Petrides KV, Mikolajczak M, Mavroveli S, Sanchez-Ruiz M-, Furnham A, Pérez-González J-. Developments in trait emotional intelligence research. Emot Rev [Internet]. 2016; 8(4): 335-41.
- [Background] Carriere JSA, Seli P, Smilek D. Wandering in both mind and body: individual differences in mind wandering and inattention predict fidgeting. Can J Exp Psychol. 2013 Mar;67(1):19-31. doi: 10.1037/a0031438. PMID 23458548
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Garzon Umerenkova A, de la Fuente Arias J, Martinez-Vicente JM, Zapata Sevillano L, Pichardo MC, Garcia-Berben AB. Validation of the Spanish Short Self-Regulation Questionnaire (SSSRQ) through Rasch Analysis. Front Psychol. 2017 Mar 1;8:276. doi: 10.3389/fpsyg.2017.00276. eCollection 2017. PMID 28298898
- [Background] Villadangos M, Errasti J, Amigo I, Jolliffe D, Garcia-Cueto E. Characteristics of Empathy in young people measured by the Spanish validation of the Basic Empathy Scale. Psicothema. 2016 Aug;28(3):323-9. doi: 10.7334/psicothema2016.6. PMID 27448268